CLINICAL TRIAL: NCT05006040
Title: Safety and Feasibility Study of a Hybrid Closed-loop Insulin Delivery System for Children and Young Adults With High Risk Acute Lymphoblastic Leukemia
Brief Title: HCL Single Arm Pilot Study in Treatment of Hyperglycemia of Pediatric ALL
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other); DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-2695.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-07-07; First posted 2021-08-16 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: High Risk Acute Lymphoblastic Leukemia

STUDY DESIGN:
Intervention Model Description: This is a non-randomized prospective cohort study about the safety and feasibility of a commercially available hybrid closed loop insulin delivery system in children and young adults with high-risk ALL who are at high risk of hyperglycemia due to an intensive chemotherapy regimen containing steroids and asparaginase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid Closed-Loop Insulin System During Chemo with Steroid and Asparaginase (Experimental): Subjects will receive insulin via hybrid closed-loop insulin delivery system during the chemotherapy phases that contains steroid and asparaginase. This treatment will be initiated within 4 days of starting induction chemotherapy treatment.
  Interventions: Device: Hybrid Closed Loop System

INTERVENTIONS:
Device: Hybrid Closed Loop System — Participants will utilize the Tandem Control-IQ Professional Hybrid Closed Loop artificial pancreas system [25, 26]. This device consists of the Dexcom G6 Continuous glucose monitor (or a more recent interoperable CGM), the Tandem t:slim X2 continuous subcutaneous insulin infusion pump, and the Control-IQ professional hybrid closed loop control algorithm. The CGM is generally replaced by parents or patients and then replaced after sensor expiration or if it falls off. This CGM, like all future iCGMs, is factory calibrated and approved for direct dosing of insulin. In addition, while the system is in use, patients will conduct blood glucose level checks at least four times a day with a fingerstick and calibrate the CGM if the measurements differ by more than 20 mg/dL of fingerstick blood glucose level. The t:slim X2 insulin pump delivers rapid acting insulin via a subcutaneous cannula which is placed by parents or patients and then replaced every 3 days [30].
  Other Names: Tandem Control-IQ Professional Hybrid Closed Loop system

SUMMARY:
The overall objective of this pilot study is to determine the safety and feasibility of a hybrid closed-loop insulin delivery system for children and young adults with high risk acute lymphoblastic leukemia, during the induction chemotherapy phase while they are exposed to steroids and asparaginase that cause hyperglycemia.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to determine the safety and feasibility of a hybrid closed-loop insulin delivery system for children and young adults with high risk acute lymphoblastic leukemia, during the induction chemotherapy phase while they are exposed to steroids and asparaginase that cause hyperglycemia. Insulin therapy would be beneficial in reducing hyperglycemia-associated complications in this period and thereby could improve other outcomes. The primary objective of the current pilot proposal is to demonstrate that hybrid closed loop pump therapy is a safe to be used in children and young adults with high risk acute lymphoblastic leukemia. If successful, the results of this study will be used to plan and support a larger, multi-center clinical trial and a grant proposal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 10 years old and above
2. Patients who are newly diagnosed with high-risk acute lymphoblastic leukemia
3. Patients who have started or will start an induction chemotherapy regimen containing steroid and asparaginase
4. Patients (if over 18 years of age) or parent/guardian (if the patient is under 18 years of age) must be fluent in reading and speaking English
5. Parent or guardian living in the home with the participant who also receives training on diabetes, CGM, HCL therapy, and the safety protocols

Exclusion Criteria:

1. Preexisting diabetes
2. Severe psychiatric disease or developmental delays, that might interfere with ability to provide informed consent
3. Active skin condition that would affect sensor placement
4. Any other medical condition which in the opinion of the investigators impairs the person's ability to safely participate in the trial, including but limited to:

   1. Significant chronic kidney disease (eGFR <60) or requiring hemodialysis
   2. Significant liver disease
   3. History of adrenal insufficiency
   4. History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
   5. History of thyroid cancer
5. Use of intravenous or oral acetaminophen more than 60 mg/kg/day (maximum 4000 mg/day)

Ages: 10 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
CGM Time in hypoglycemia (blood glucose < 70 mg/dL) | 35 days
  The primary outcome measures for this study will be the safety of HCL insulin delivery by hypoglycemia exposure. One of the primary endpoints is CGM Time in hypoglycemia (defined as blood glucose < 70 mg/dL).
Number of episodes of symptomatic hypoglycemia | 35 days
  The primary outcome measures for this study will be the safety of HCL insulin delivery by hypoglycemia exposure. One of the primary endpoints is the number of episodes of symptomatic hypoglycemia. At each study visit, subjects will be asked about symptoms, such as shakiness, dizziness, blurred/impaired vision, sweating, pallor, clumsiness, difficulty paying attention, tingling around the lips, tongue or cheeks, change in mental status, or seizure.
Rate of infection at the CGM insertion site | 35 days
  Rate of infection at the CGM insertion site, measured in occurrences per patient-day.
Rate of bleeding at the CGM insertion site | 35 days
  Rate of bleeding at the CGM insertion site, measured in occurrence per patient-day.
Rate of infection at the HCL insulin infusion site | 35 days
  Rate of infection at the HCL insulin infusion site, measured in occurrence per patient-day.
Rate of bleeding at the HCL insulin infusion site | 35 days
  Rate of bleeding at the HCL insulin infusion site, measured in occurrence per patient-day.

SECONDARY OUTCOMES:
Efficacy of glycemic control with HCL insulin delivery assessed by Time in Ranges (TIR) | 35 days
  Time in Ranges (TIRs) refers to percent of the time spent in a specific range of blood glucose levels, adding valuable information to assess the level of glycemic control. Usually a range of 70-180 mg/dL is used, but occasionally a more stringent 70-140 mg/dL is used. In this study, we will obtain %CGM TIRs in both ranges.
Efficacy of glycemic control with HCL insulin delivery assessed by mean sensor glucose level | 35 days
  Mean glucose level will be obtained from CGM data to evaluate for glycemic variability
Rate of infection in episodes per patient-days | 35 days
  Rate of infection, length of hospitalization, length of PICU admission, rate of remission at the end of induction, and need for re-admission will be obtained as a part of clinical outcomes. These outcomes will be compared to a historical control group to investigate the effect size of relationships between glycemic control and clinical outcome. This exploratory aim will investigate correlations between glycemic control and outcomes to determine effect sizes for future studies and grant proposals.
Length of hospitalization in days per patient | 35 days
  Rate of infection, length of hospitalization, length of PICU admission, rate of remission at the end of induction, and need for re-admission will be obtained as a part of clinical outcomes. These outcomes will be compared to a historical control group to investigate the effect size of relationships between glycemic control and clinical outcome. This exploratory aim will investigate correlations between glycemic control and outcomes to determine effect sizes for future studies and grant proposals.
Length of PICU admission in days per patient | 35 days
  Rate of infection, length of hospitalization, length of PICU admission, rate of remission at the end of induction, and need for re-admission will be obtained as a part of clinical outcomes. These outcomes will be compared to a historical control group to investigate the effect size of relationships between glycemic control and clinical outcome. This exploratory aim will investigate correlations between glycemic control and outcomes to determine effect sizes for future studies and grant proposals.
Rate of remission at the end of induction in percent | 35 days
  Rate of infection, length of hospitalization, length of PICU admission, rate of remission at the end of induction, and need for re-admission will be obtained as a part of clinical outcomes. These outcomes will be compared to a historical control group to investigate the effect size of relationships between glycemic control and clinical outcome. This exploratory aim will investigate correlations between glycemic control and outcomes to determine effect sizes for future studies and grant proposals.
Need for readmission during the induction phase in percent | 35 days
  Rate of infection, length of hospitalization, length of PICU admission, rate of remission at the end of induction, and need for re-admission will be obtained as a part of clinical outcomes. These outcomes will be compared to a historical control group to investigate the effect size of relationships between glycemic control and clinical outcome. This exploratory aim will investigate correlations between glycemic control and outcomes to determine effect sizes for future studies and grant proposals.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Forlenza, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No